CLINICAL TRIAL: NCT06223399
Title: Randomized Controlled Trial Comparing Imaging-based Programming With Threshold-assessment Based Programming of Deep Brain Stimulation for Parkinson's Disease
Brief Title: DBS Imaging-based vs. Threshold Assessment-based Programming
Acronym: DBS-ITAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Rob M.A. de Bie, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL84601.018.23
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Deep Brain Stimulation; Parkinson Disease; Imaging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study will be a mono center prospective randomized open label blinded endpoint (PROBE) design trial comparing imaging-based DBS programming with DBS programming based on threshold assessment.
Who Masked: Outcomes Assessor
Masking Description: Patients cannot be blinded for the treatment allocation, because the person who programs the DBS receives either dictated stimulation parameters based on imaging or proceeds with care as usual with the threshold assessment. Blinded assessment of the primary outcome will be done by means of a physical examination blinded for randomization arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaging-based (Experimental): 66 patients with Parkinson's disease will receive imaging-based DBS programming
  Interventions: Other: Imaging-based programming
- Threshold assessment-based (Active Comparator): 66 patients with Parkinson's disease will receive DBS programming based on the threshold assessment
  Interventions: Other: Threshold assessment-based programming

INTERVENTIONS:
Other: Imaging-based programming — Preferred contact point(s) and settings for DBS programming will be determined based on the visualization of the electrodes in the patient-specific anatomy and the volume of tissue activated (VTA; i.e., the tissue enclosed within an iso-surface of the activation function). This will be determined with help of the software program Brainlab with the GUIDE XT module.
  Arms: Imaging-based
Other: Threshold assessment-based programming — The preferred contact point(s) and settings for DBS programming will be determined according to current clinical practice. During the threshold assessment, the amount of electrical current needed to generate symptomatic improvement and the amount of electrical current needed to generate adverse-effects are determined for every contact point of both DBS leads by increasing current with 0.5 mA steps from 0 to approximately 5.0 mA. With each step, severity of Parkinson symptoms and presence of possible adverse-effects are assessed. For each side (i.e., left and right), the contact point with the most favorable trade-off between clinical improvement and adverse effects will be used for stimulation.
  Arms: Threshold assessment-based

SUMMARY:
The goal of this single-center prospective, randomized, open-label clinical trial is to compare the effectiveness of imaging-based DBS programming with threshold assessment-based DBS programming in patients with Parkinson's disease and motor response fluctuations.

The main question the study aims to answer is:

Is the improvement of motor symptoms in the OFF-drug phase following STN DBS for Parkinson's disease, using imaging-based DBS programming only, non-inferior to the improvement of motor symptoms following DBS programming with threshold assessment at six months follow-up?

Participants will be randomized to imaging-based programming or to threshold assessment-based programming. The main clinical outcome is motor symptoms; secondary outcomes are level of physical disability and quality of life, among others.

DETAILED DESCRIPTION:
Rationale:

Deep Brain Stimulation (DBS) of the subthalamic nucleus (STN) is an established treatment for disabling motor symptoms of Parkinson's disease (PD). Correct programming of DBS settings to provide optimal stimulation within the target region is crucial for a successful clinical outcome. To date, programming DBS settings is based on the selection of contact point(s) and stimulation parameters with standardized threshold assessments: for each contact point the current is increased in small steps and the severity of motor symptoms and possible adverse effects are assessed with each step. This process is challenging and time consuming because of the vast number of possible parameter combinations. Furthermore, individual variation in patient anatomy, placement of DBS leads and the occurrence of adverse effects must be considered. This results in long programming sessions that can be exhausting for patients and often leads to inconclusive results due to fatigue. Imaging techniques have been improved greatly over the years and could be useful for programming of DBS settings based on patient-specific anatomy.

Objective:

The aim of this study is to determine whether imaging-based DBS programming for the treatment of Parkinson's motor symptoms in STN DBS is non-inferior to the current standard practice of clinical threshold assessment-based DBS programming.

Study design:

The study is a single-center prospective, randomized, open-label, blinded end-point (PROBE design) clinical trial. Following surgery for DBS implantation, in total 132 patients will be randomized in a 1:1 ratio to initial imaging-based DBS programming (Imaging group) or to DBS programming based on initial threshold assessment (Threshold group). Follow-up is six months and consists of 3 study visits.

Study population:

Patients are eligible for the trial if they will have bilateral STN DBS for Parkinson motor symptoms at Amsterdam UMC.

Interventions:

In both groups (i.e., Imaging and Threshold), DBS programming will start two to three weeks after DBS surgery. For the DBS programming patients are admitted in the hospital for a day while they are off Parkinson medication.

Imaging group:

With the use imaging investigators are capable to visualize the location of the DBS lead within the individual's segmented anatomy and volume of tissue activated (VTA; i.e., the tissue enclosed within an iso-surface of the activation function), this may have the potential to improve programming of the stimulation parameters and outcomes. For this, the postoperative CT-scan is used to localize the DBS leads and the surrounding anatomic structures are reconstructed with the patient's preoperative MRI scan. Based on the patient-specific anatomy the DBS settings (appropriate contacts, amplitude, and pulse width) can be determined that produce the ideal VTA within the target and minimalizing stimulation of the surrounding structures. These settings can then be used as starting point for the programming of the stimulation parameters.

Threshold group:

Each DBS-electrode has four to 16 contact points, close to the tip, from where electrical current can be emitted. When programming DBS, the contact point or combination of contact points used for stimulation and the optimal electrical stimulation parameters are chosen. Two to three weeks after the surgery the clinician turns on the DBS. For this purpose, the patient is admitted to the hospital, and the initial threshold assessment is performed for each contact point. A crucial step in this process is to determine for each separate contact point, the amount of current needed to generate symptomatic improvement and the amount of current that generates adverse effects. To determine these thresholds, current is increased with 0.5 milliampere (mA) steps from 0 to approximately 5.0 mA, sequentially for each contact point, and the severity of Parkinson symptoms and possible adverse effects are assessed with each step. For this threshold-assessment, patients have to be off Parkinson medication (OFF-drug phase). Based on the threshold-assessments the active contact point(s) and stimulation parameters are selected. The DBS current is usually gradually increased over weeks to months with corresponding adjustments of the pharmacological treatment. For patients with bilateral DBS and four contact points on each electrode, the threshold-assessment takes about three hours.

The patient has a 50% chance of being randomized to initial imaging-based DBS programming (i.e., Imaging group). The expected benefit for this group is that they will not need the threshold-assessment and therefore have less burden due to less hospital visits for the programming. There are no extra risks associated with participation in this study. If the stimulation parameters found with imaging-based programming only do not yield enough effect in the Imaging group, the healthcare professionals can choose to execute the threshold-assessment for these patients.

Impact:

The results of the study may well contribute to reducing the burden of DBS treatment. If imaging-based programming is non-inferior to threshold assessment-based programming, this may result in more efficient programming sessions with reduced programming time (less use of health-care resources) and less discomfort for patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosis based on the clinical diagnostic criteria of Movement Disorder Society
* Scheduled for DBS screening
* Age of 18 years or older
* Understand the Dutch language

Exclusion Criteria:

* Legally incompetent adults
* No written informed consent
* Previous functional stereotactic neurosurgery
* Dementia
* Current depression or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III in OFF phase | Change from baseline to 6 months of DBS.
  The MDS-UPDRS III measures severity of Parkinson's disease. The scores range between 0 - 132, higher scores indicating worse motor symptoms.

SECONDARY OUTCOMES:
MDS-UPDRS III in ON phase | Change from baseline to 6 months of DBS.
  The MDS-UPDRS III measures severity of Parkinson's disease. The scores range between 0 - 132, higher scores indicating worse motor symptoms.
MDS-UPDRS IV | Change from baseline to 6 months of DBS.
  Part IV of the MDS-UPDRS evaluates two motor complications: dyskinesia duration and severity and motor fluctuations by means of six questions administered by a healthcare professional. The fourth part ranges from 0 to 24, with a higher score indicating greater disability.
MDS-UPDRS I | Change from baseline to 6 months of DBS.
  Part I of the MDS-UPDRS evaluates the non-motor impact on patients' experiences of daily living by means of questions administered by a healthcare professional and self-administered questions. The first part ranges from 0 to 52, with a higher score indicating greater disability.
MDS-UPDRS II in ON phase | Change from baseline to 6 months of DBS.
  Part II of the MDS-UPDRS evaluates motor experiences in daily living by means of a self-administered questionnaire. The second part ranges from 0 to 52 with a higher score indicating greater disability.
Academic Medical Center Linear Disability Score (ALDS) | Change from baseline to 6 months of DBS.
  The ALDS measures the disability status of patients with a broad range of diseases. It is expressed by the ability to perform activities in daily living and each item is scored separately. The scores range between 0 - 100, lower scores indicating more disability.
Parkinson's Disease Questionnaire 39 (PDQ-39) | Change from baseline to 6 months of DBS.
  The PDQ-39 evaluates the quality of life by means of a questionnaire containing 39 items and eight dimensions (i.e., mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort). The total score is the sum of the eight different dimensions and yields a score between 0 and 100. A higher score indicates less quality of life.
Patient satisfaction of the outcome of treatment | At 6 months of DBS
  The degree of satisfaction scored by the patient on a 5-point Likert scale, with higher scores indicating higher experienced satisfaction.
Patient evaluation of the burden of therapy | At 6 months of DBS
  The degree of experienced burden scored by the patient on a 5-point Likert scale, with higher scores indicating higher experienced burden.
Adverse effects | At 6 months of DBS
  Number and sort of adverse effects observed during six months follow-up after DBS.
Use of care | At 6 months of DBS
  Total contact moments (via telephone or in hospital) during six months follow-up after DBS.
Total duration of programming sessions | At 6 months of DBS
  Combined duration of programming sessions during the follow-up period after DBS.
Final DBS settings | At 6 months of DBS
  Final stimulation parameters at 6 months after follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rob de Bie, Prof, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in the publication will be made available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It will be made available one year after the last study visit of the last participant
Access Criteria: Upon request